CLINICAL TRIAL: NCT02070081
Title: Patient Profiling for Successful Weight Loss After Gastric Bypass or Sleeve Surgery
Brief Title: Weight Loss Following Gastric Bypass or Sleeve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Bariatric Clinic, Department of Surgery, Køge Hospital, Denmark (Unknown); Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Arne Astrup, Prof., MD, Head of Department of Nutrition, Exercise and Sports, University of Copenhagen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO Bypass
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Experimental)
  Interventions: Procedure: Roux-en-Y gastric bypass surgery or sleeve surgery

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass surgery or sleeve surgery

SUMMARY:
The overall aim is to study the multiple factors determining the variation of weight loss after Roux-en-Y Gastric Bypass (RYGB) and Sleeve surgery.

The specific aims are to evaluate:

a) what explains the large individual differences in weight loss seen after RYGB and Sleeve surgery, b) if it is possible pre-operatively to identify which patients will not obtain beneficial effects of bariatric surgery in relation to weight loss and quality of life and c) if patients in need of improved care can be identified pre- and/or early post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* All patients approved for bariatric surgery at Bariatric Clinic, Køge Hospital, Denmark

Exclusion Criteria:

* Inability to comply with the study protocol

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Weight loss | 3 month preoperatively, 1 week preoperatively, 6 weeks postoperatively, 6 month postoperatively and 18 month postoperatively

SECONDARY OUTCOMES:
Metabolic profile | 3 month preoperatively, 1 week preoperatively, 6 month postoperatively and 18 month postoperatively
  Insulin, glucose, C-peptide, GIP, glucagon, TSH, thyroid hormones, vitamin D and blood lipids
Physical activity | 3 month preoperatively, 1 week preoperatively, 6 month postoperatively and 18 month postoperatively
Appetite sensation | 3 month preoperatively, 1 week preoperatively, 6 weeks postoperatively, 6 month postoperatively and 18 month postoperatively
  Following a test meal with the use of visual analogue scales (VAS)
Taste preferences and taste perception | 3 month preoperatively, 1 week preoperatively, 6 weeks postoperatively, 6 month postoperatively and 18 month postoperatively
  Sensory tests, picture displays (all visits) and an ad libitum test meals (3 months preoperatively and 6 months postoperatively) are used to investigate changes in taste and food preferences (liking and wanting) and taste perception
Mental health | 3 month preoperatively, 6 month postoperatively and 18 month postoperatively
Social resources | 3 month preoperatively, 1 week preoperatively, 6 weeks postoperatively, 6 month postoperatively and 18 month postoperatively
Gut microbiota | 1 week preoperatively, 6 month postoperatively
Appetite-regulating hormones | 3 month preoperatively, 1 week preoperatively, 6 month postoperatively and 18 month postoperatively
  GLP-1, PYY, leptin, ghrelin, OXM, CCK, glicentin
Bile acids and fibroblast growth factors | 3 month preoperatively, 1 week preoperatively, 6 month postoperatively and 18 month postoperatively
Genetics | 3 month preoperatively
Body composition | 3 month preoperatively, 1 week preoperatively, 6 weeks postoperatively, 6 month postoperatively and 18 month postoperatively
  By DXA scans
Cortisol | 3 month preoperatively and 18 month postoperatively
  Measured in hair
Neural activity in reward-processing brain centers | preoperatively and 6 month postoperatively
  By functional magnetic resonance imaging (fmri)
Rewarding value of food | preoperatively and 6 month postoperatively
  Behavioral test

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Science, NEXS, Frederiksberg, Denmark

REFERENCES:
- [Derived] Nielsen MS, Ritz C, Wewer Albrechtsen NJ, Holst JJ, le Roux CW, Sjodin A. Oxyntomodulin and Glicentin May Predict the Effect of Bariatric Surgery on Food Preferences and Weight Loss. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgaa061. doi: 10.1210/clinem/dgaa061. PMID 32016415
- [Derived] Nielsen MS, Andersen INSK, Lange B, Ritz C, le Roux CW, Schmidt JB, Sjodin A, Bredie WLP. Bariatric Surgery Leads to Short-Term Effects on Sweet Taste Sensitivity and Hedonic Evaluation of Fatty Food Stimuli. Obesity (Silver Spring). 2019 Nov;27(11):1796-1804. doi: 10.1002/oby.22589. Epub 2019 Sep 26. PMID 31556242
- [Derived] Taekker L, Lunn S. The effect of mental health on weight loss after bariatric surgery. Dan Med J. 2019 Feb;66(2):A5532. PMID 30722827
- [Derived] Sondergaard Nielsen M, Rasmussen S, Just Christensen B, Ritz C, le Roux CW, Berg Schmidt J, Sjodin A. Bariatric Surgery Does Not Affect Food Preferences, but Individual Changes in Food Preferences May Predict Weight Loss. Obesity (Silver Spring). 2018 Dec;26(12):1879-1887. doi: 10.1002/oby.22272. Epub 2018 Nov 13. PMID 30421858
- [Derived] Christensen BJ, Schmidt JB, Nielsen MS, Taekker L, Holm L, Lunn S, Bredie WLP, Ritz C, Holst JJ, Hansen T, Hilbert A, le Roux CW, Hulme OJ, Siebner H, Morville T, Naver L, Floyd AK, Sjodin A. Patient profiling for success after weight loss surgery (GO Bypass study): An interdisciplinary study protocol. Contemp Clin Trials Commun. 2018 Feb 17;10:121-130. doi: 10.1016/j.conctc.2018.02.002. eCollection 2018 Jun. PMID 30023446
- [Derived] Nielsen MS, Christensen BJ, Ritz C, Rasmussen S, Hansen TT, Bredie WLP, le Roux CW, Sjodin A, Schmidt JB. Roux-En-Y Gastric Bypass and Sleeve Gastrectomy Does Not Affect Food Preferences When Assessed by an Ad libitum Buffet Meal. Obes Surg. 2017 Oct;27(10):2599-2605. doi: 10.1007/s11695-017-2678-6. PMID 28411313